CLINICAL TRIAL: NCT01231529
Title: A Phase I, Open-Label, Parallel-Group, Two-Part, Adaptive Study to Evaluate the Pharmacokinetics and Safety of GSK1349572 in Subjects With Hepatic Impairment and Healthy Matched Control Subjects (ING113097)
Brief Title: GSK1349572 Hepatic Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 113097; NCT01377714 (obsolete NCT alias)
Record Dates: First submitted 2010-10-14; First posted 2010-11-01 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Healthy Subjects; Hepatic Impairment; Infection, Human Immunodeficiency Virus; HIV Infections
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 Cohort 1 (Experimental): 8 subjects with moderate hepatic impairment defined by a Child-Pugh score of 7 to 9 will receive a single oral dose of GSK1349572 50 mg in the morning followed by 72 hour serial PK sampling. There will be a screening visit within 30 days prior to the dose of study drug and a follow-up visit within 7-10 days after the study drug.
  Interventions: Drug: GSK1349572
- Part 1 Cohort 2 (Experimental): 8 healthy subjects matched by gender, age and BMI to the subjects in Cohort 1 will receive a single oral dose of GSK1349572 50 mg in the morning followed by 72 hour serial PK sampling. There will be a screening visit within 30 days prior to the dose of study drug and a follow-up visit within 7-10 days after the study drug.
  Interventions: Drug: GSK1349572
- Part 2 Cohort 3 (Experimental): 8 subjects with mild hepatic impairment defined by a Child-Pugh score of 5 to 6 will receive a single oral dose of GSK1349572 50 mg in the morning followed by 72 hour serial PK sampling. There will be a screening visit within 30 days prior to the dose of study drug and a follow-up visit within 7-10 days after the study drug. This cohort will only be done if the AUC from Cohort 1 is greater than or equal to 2 times the AUC from Cohort 2.
  Interventions: Drug: GSK1349572
- Part 2 Cohort 4 (Experimental): 8 healthy subjects matched by gender, age and BMI to the subjects in Cohort 3 will receive a single oral dose of GSK1349572 50 mg in the morning followed by 72 hour serial PK sampling. There will be a screening visit within 30 days prior to the dose of study drug and a follow-up visit within 7-10 days after the study drug. This cohort will only be done if the AUC from Cohort 1 is greater than or equal to 2 times the AUC from Cohort 2.
  Interventions: Drug: GSK1349572

INTERVENTIONS:
Drug: GSK1349572 — All subjects will receive a single dose of GSK1349572 50 mg. GSK1349572 is an experimental drug in the integrase inhibitor class being developed for the treatment of HIV infection. GSK1349572 is not approved by the FDA.

SUMMARY:
GSK1349572 is an integrase inhibitor that is currently in clinical development for the treatment of human immunodeficiency virus (HIV) infection. GSK1349572 is metabolized primarily by uridine diphosphate glucuronosyltransferase (UGT)1A1 with a minor role of Cytochrome P450 (CYP)3A. Hepatic impairment could potentially alter the clearance and plasma protein binding of GSK1349572. This study will evaluate the single dose pharmacokinetics and safety of GSK1349572 in healthy subjects and in subjects with mild or moderate hepatic impairment based on Child-Pugh category.

This is a single-dose, open-label, parallel group, two-part, adaptive study in adult males and females with mild or moderate hepatic impairment and matched, healthy control subjects with normal hepatic function. Healthy control subjects (16) will be matched for gender, age, and BMI to the subjects in the mild (8) or moderate (8) hepatic impairment category. In Part 1, approximately 8 subjects with moderate hepatic impairment (cohort 1) and 8 matched, control subjects (cohort 2) will each receive GSK1349572 50 mg as a single dose in the fasted state followed by pharmacokinetic sampling for total concentrations of GSK1349572 in plasma. Free (unbound) plasma concentrations of GSK1349572 will also be evaluated at sparse, selected time points. If the geometric mean total plasma area under the concentration curve (AUC) of GSK1349572 is increased by > 2-fold in moderately impaired subjects compared to matched controls, Part 2 will be conducted to evaluate GSK1349572 pharmacokinetics in another group of subjects with mild impairment (8, cohort 3) and matched, control subjects (8, cohort 4). Vital signs, electrocardiograms (ECGs), and adverse events will be monitored throughout the study. A follow-up visit will occur 7-10 days after the dose of study drug.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* A male or female is eligible for study participation if he/she: Is healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.

OR (Part 1 subjects only) Is considered to have moderate hepatic insufficiency (of any etiology) and has been clinically stable for at least 1 month prior to screening. To be classified as having moderate hepatic insufficiency, subjects must have: A Child-Pugh score of 7-9 and previous confirmation of liver cirrhosis by liver biopsy or other medical imaging technique (including laparoscopy, computed tomography (CT) scan, magnetic resonance imaging (MRI) or ultrasonography) associated with an unambiguous medical history (such as evidence of portal hypertension) OR (Part 2 subjects only) Is considered to have mild hepatic insufficiency (of any etiology) and has been clinically stable for at least 1 month prior to screening. To be classified as having mild hepatic insufficiency, subjects must have: A Child-Pugh score of 5-6 and previous confirmation of liver cirrhosis by liver biopsy or other medical imaging technique (including laparoscopy, CT scan, MRI or ultrasonography) associated with an unambiguous medical history (such as evidence of portal hypertension).

* Aged between 18 and and 70 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory] or Child-bearing potential and agrees to use one of the contraception methods listed for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 3 days after the last dose of study medication.
* Body weight greater than or equal to 50 kg for men and women and body mass index (BMI) within the range 19- 41 kg/m2 for hepatically impaired subjects; healthy matched control subjects will be matched to BMI +/- 20% and must also remain in the BMI range of 19- 41 kg/m2.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

A healthy subject will not be eligible for inclusion in this study if any of the following criteria apply:

* A positive Hepatitis B surface antigen or positive Hepatitis C antibody result at screening.
* A positive test for HIV antibody at screening.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* If heparin is used during pharmacokinetic (PK) sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy and inflammatory bowel disease should be excluded. Subjects with a history of peptic ulceration or pancreatitis within the preceding 6 months of screening should be excluded.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of regular use of tobacco or nicotine-containing products within 3 months prior to screening.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5x upper limit of normal (ULN); alkaline phosphatase or bilirubin ≥ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of Gilbert's disease.
* The subject's systolic blood pressure is outside the range of 90-145mmHg, or diastolic blood pressure is outside the range of 45-95mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination) per protocol

A subject with mild or moderate hepatic impairment will not be eligible for inclusion in this study if any of the following criteria apply:

* Evidence of recent infection with Hepatitis B and/or Hepatitis C within preceding 6 months. Subjects with chronic Hepatitis B or C (duration>6 months) are eligible for enrolment.
* A positive test for HIV antibody at screening.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines. A positive drug screen will be allowed if it is due to a prescribed medication.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Subjects with a pre-existing condition (except hepatic impairment) interfering with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy and inflammatory bowel disease should be excluded. Subjects with a history of peptic ulceration or pancreatitis within the preceding 6 months of screening should be excluded. Subjects with previous gastrointestinal (GI) surgery (except appendectomy or gall bladder removal more than three months prior to study) should be excluded.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects using any concurrent prohibited medication. Use of common medications which are permitted during the study are listed in the protocol (permitted medications).
* Subjects receiving lactulose who are medically unable to halt lactulose administration from 8h before dosing with study drug to 4h after dosing with study drug.
* Subjects with a change in dose regimen of medically required medication within the 2 weeks prior to dosing.
* Subjects with fluctuating or rapidly deteriorating hepatic function. Assessment of the stability of the subject's hepatic function will be determined by the investigator.
* Subjects with creatinine clearance less than or equal to 50 mL/min (calculated by the Cockcroft-Gault Formula).
* Subjects with advanced ascites (Grade 3).
* Subjects whose serum sodium levels are less than or equal to 125 mmol/L.
* Subjects whose platelets are less than 50,000 x 109/L of blood.
* Subjects with refractory encephalopathy as judged by the investigator or significant Central Nervous System (CNS) disease (e.g. dementia, or seizures) which the investigator considers will interfere with the informed consent, conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Subjects with signs of active infection.
* Subjects with esophageal variceal bleeding within the past 6 months.
* Subjects with Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement.
* Subjects with any other medical condition which, in the judgement of the investigator and medical monitor, could jeopardize the integrity of the data derived from that subject or the safety of the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11-19 (Actual); Primary Completion 2011-06-04 (Actual); Study Completion 2011-06-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC(0-t)) | 72 hours
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity),) | 72 hours
Maximum observed concentration (Cmax) | 72 hours
Concentration at 24 hours post dose (C24) | 24 hours
apparent terminal phase half-life (t1/2) | 72 hours
apparent clearance (CL/F) following oral dosing | 72 hours
Apparent volume of distribution after extravascular (e.g., oral) administration (Vz/F) | 72 hours

SECONDARY OUTCOMES:
Number of subjects with adverse events | 72 hours
Unbound concentration in plasma of GSK1349572 at 3 hours post dose | 3 hours
Time of occurrence of Cmax (tmax) | 24 hours
Number of subjects using concurrent medications | 72 hours
Change from baseline in clinical laboratory tests | 72 hours
Change from baseline in vital signs | 3 hours
Unbound concentration in plasma of GSK1349572 at 24 hours post dose | 24 hours
Unbound fraction in plasma of GSK1349572 at 3 hours post dose | 3 hours
Unbound fraction in plasma of GSK1349572 at 24 hours post dose | 24 hours
Lag time before observation of drug concentrations in sampled matrix (tlag) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Song IH, Borland J, Savina PM, Chen S, Patel P, Wajima T, Peppercorn AF, Piscitelli SC. Pharmacokinetics of Single-Dose Dolutegravir in HIV-Seronegative Subjects With Moderate Hepatic Impairment Compared to Healthy Matched Controls. Clin Pharmacol Drug Dev. 2013 Oct;2(4):342-348. doi: 10.1002/cpdd.55. Epub 2013 Aug 16. PMID 26097786